CLINICAL TRIAL: NCT04775212
Title: Effects of Desflurane and Sevoflurane Anesthesia on Postoperative Liver Functions in Pediatric Cancer Patients With Elevated Liver Enzymes
Brief Title: Desflurane and Sevoflurane in Pediatrics With Elevated Liver Enzymes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Norma Osama Abdalla Zayed, assistant lecturer, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AP2101-50101
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Liver Functions Tests
Keywords: Desflurane,Sevoflurane,liver enzymes,cancer
MeSH Terms: interventions — Desflurane; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- desflurane (Active Comparator): patients to be anesthetized with desflurane
  Interventions: Drug: Desﬂurane
- sevoflurane (Active Comparator): patients to be anesthetized with sevoflurane
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Desﬂurane — compare effects of inhaled anaesthetic desflurane and sevoflurane on liver functions.
  Other Names: Suprane
  Arms: desflurane
Drug: Sevoflurane — Sevoflurane
  Arms: sevoflurane

SUMMARY:
It is designed to compare effects of inhaled anaesthetic desflurane and sevoflurane on liver functions in pediatric cancer patients

DETAILED DESCRIPTION:
Patients will be randomly allocated into two groups using a sealed envelope technique: desflurane group (Des group, n = 30) and sevoflurane group (sevo group, n = 30).

Anesthesia monitoring included electrocardiogram, continuous arterial and pulse oximetry, capnography, urine output, nerve stimulator, and esophageal core temperature.

Anesthesia will be induced with Propofol 2 mg/kg ,FentanyL 2 μg/kg and atracurium (0.5 mg/kg) was administered to achieve muscle relaxation before endotracheal intubation. End-tidal desflurane or sevoflurane concentrations during the induction were limited to 2 minimal alveolar concentration (MAC). Concentrations of inhalational anesthetics were measured using an anesthetic gas analyser (Datex-Ohmeda, Helsinki, Finland). For the maintenance of anesthesia, the inspired desflurane or sevoflurane concentration was carefully titrated to maintain the end-tidal concentration of 1 MAC. A constant fresh gas flow of 3 l/min (medical-grade air in oxygen to make inspiratory oxygen fraction 0.5) was used during the maintenance of anesthesia. Ventilation was controlled with a tidal volume of 7-10 ml/kg and ventilatory rate was adjusted to maintain an end tidal carbon dioxide ( CO2 )of 35-40 mmHg. to maintain intraoperative blood pressure (BP) and heart rate (HR) within 20% of preoperative values. additional Atracurium will be administered as appropriate. Nerve stimulator was used to monitor neuromuscular blockade on the right adductor pollicis. Hypotension (a drop in systolic BP to the extent of 30% or more or the systolic BP being less than the preoperative values) was treated with volume replacement and, when necessary, with intravenous ephedrine in incremental doses .Bradycardia (HR < 50 beats per min) was treated with atropine if needed.

Aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin (TB), prothrombin time (PT) expressed in international normalized ratio (INR), albumin, platelet count (PLT), and hemoglobin (Hb) were analysed at preoperative period, immediately after operation, and on the 1st, 2nd, 3rd, 5th and 7th, postoperative days (PODs).

ELIGIBILITY:
Inclusion Criteria:

* Age >1 year and < 12 years old.
* Estimated time of surgeries within 1-3 hours.
* Elevated liver enzymes less than triple folds.

Exclusion Criteria:

* Patient refusal.
* Hepatitis positive patients.
* Raising liver enzymes.
* Hepatic surgeries.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — 2-18 years old
Enrollment: 60 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2021-10-17 (Estimated); Study Completion 2021-10-17 (Estimated)

PRIMARY OUTCOMES:
liver function test | 6 months
  measuring Aspartate aminotransferase (AST)
ALT | 6 months
  measuring alanine aminotransferase (ALT)
Total bilirubin | 6 months
  measuring total bilirubin (TB)
prothrombin time | 6 months
  measuring prothrombin time (PT) expressed in international normalized ratio (INR)
Albumin | 6 months
  measuring level of albumin.

CONTACTS AND LOCATIONS:
Overall Officials: Suzan Adlan, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National cancer institute, Cairo, Egypt